CLINICAL TRIAL: NCT05557162
Title: Artificial Intelligence Enhanced ECG to Detect Cardiac Amyloidosis: Protocol for a Pragmatic Cluster Randomized Clinical Trial (PREDICT-AMY)
Brief Title: Artificial Intelligence Enhanced ECG to Detect Cardiac Amyloidosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PREDICT-AMY; NCI-2024-00928 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PREDICT-AMY (Other: Sponsor Protocol Number); 22-005311 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-09-16; First posted 2022-09-27 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Notification of the AI ECG algorithm and the A3E scores (Experimental): Provider-facing recommendation report that alerts to provider for positive AI ECG Amyloid Score, standardized amyloid order set, diagnostic algorithm and reminders
  Interventions: Other: AI ECG Amyloid algorithm
- Usual Care (No Intervention): No alerts to provider for positive AI ECG Amyloid Score, standardized amyloid order set, diagnostic algorithm and reminders

INTERVENTIONS:
Other: AI ECG Amyloid algorithm — Artificial intelligence enabled electrocardiogram screening tool used to identify the predictive model that best differentiates those at greatest risk for an amyloidosis diagnosis
  Arms: Notification of the AI ECG algorithm and the A3E scores

SUMMARY:
The purpose of this study is to assess a novel artificial intelligence (AI)-enabled electrocardiogram (ECG)-based screening tool for improving the diagnosis of cardiac amyloidosis (CA).

DETAILED DESCRIPTION:
This pragmatic trial will be the first study to prospectively evaluate the use of the AI ECG dashboard along with an augmented report in everyday practice. The findings will also guide future implementation strategies and inform the translation of many of the current and future AI algorithms into the clinical setting. The participants are the providers. Basic demographic information about the providers will be collected as well as their reactions to the trial based educational guidance supplied to them. Patient health information will be collected on their patients using a HIPPA waiver. There will be no patient contact.

ELIGIBILITY:
Inclusion Criteria:

* Mayo Clinic cardiology or hematology providers who care for adult patients
* Mayo Clinic providers who consent to participate on this study

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20143 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To determine if AI ECG algorithm and enhanced algorithms and education enable earlier diagnosis of cardiac amyloidosisProtocol for a Pragmatic Cluster Randomized Clinical Trial (PREDICT-AMY) | 1 year
  The number of patients diagnosed with cardiac amyloidosis in cardiology and hematology practices will be compared between those providers undergoing the AI ECG intervention to those randomized to standard practice arm

SECONDARY OUTCOMES:
To determine if AI ECG and enhanced algorithms and education enable earlier diagnosis of cardiac amyloidosis intervention across different practice types (strata) | 1 year
  Performance of AI ECG intervention across cardiology and hematology practices and between community and tertiary facilities will be analyzed by measuring rates of cardiac amyloidosis diagnosis across these strata
To assess provider satisfaction with the AI ECG intervention | 1 year
  For a screening tool to be effective, it has to be user friendly. The providers randomized to the AI ECG intervention arm will be surveyed to understand their experience. This endpoint will be descriptive. Providers will answer a 6 question using a 5-point Likert scale (higher number is more favorable).
To assess differential costs between the intervention arm and the standard of care arm | 1 year
  Upon trial completion, the difference in clinical expenditures between the intervention and standard of care arms will be compared. To this end, the rates of test ordering will be counted and compared between the interventional arm and the standard of care arm. A cost will be assigned to each test to calculate expenditures per correct diagnosis. The test of interest will include: NT-proBNP, troponin, protein electrophoresis with isotyping, serum immunoglobulin free light chains, 24-hour urinary protein with immunofixation, cardiac magnetic resonance imaging, echocardiogram, technetium pyrophosphate nuclear cardiac scintigraphy , endomyocardial biopsy, and fat aspirate.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Dispenzieri, MD, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic Health System - Eau Claire, Eau Claire, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials